CLINICAL TRIAL: NCT03160586
Title: Stuttering Severity and Anxiety in Egyptian School-age Children
Brief Title: Stuttering and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Abdelraheem, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SSI
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Stuttering, Childhood; Anxiety Disorders
Keywords: Stuttering; Anxiety
MeSH Terms: conditions — Stuttering; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stutter (Active Comparator): Children who stuttering
  Interventions: Diagnostic Test: Stuttering severity instrument-3; Diagnostic Test: Child Behavior Checklist for age 4-18
- Control (Active Comparator): Children who non stuttering
  Interventions: Diagnostic Test: Child Behavior Checklist for age 4-18

INTERVENTIONS:
Diagnostic Test: Stuttering severity instrument-3 — To measure of degree of stuttering in child
  Arms: Stutter
Diagnostic Test: Child Behavior Checklist for age 4-18 — To measure of percent of anxiety in child by ask parents about his or her behaviour

SUMMARY:
Stuttering was defined as a common neurodevelopmental speech disorder characterized by repetitions, prolongations, and interruptions in the flow of speech. In other words, stuttering is a speech disorder characterized by involuntary disruptions to speech which impede the capacity to communicate effectively.

Physiological and emotional anxiety has been reported in persons who stutter. It has been reported that as high as 44% of clients seeking treatment for stuttering could be assigned a co-occurring social phobia or social anxiety diagnosis.

DETAILED DESCRIPTION:
According to the Diagnostic and Statistical Manual of Mental Disorders, social anxiety disorder is characterized by marked or intense fear of social or performance-based situations where scrutiny or evaluation by others may occur. Feared situations often include speaking in public, meeting new people, and talking with authority figures.

There are several reasons to expect that stuttering may be associated with social anxiety disorder. To begin with, stuttering is accompanied by numerous negative consequences across the lifespan which may increase vulnerability to social and psychological difficulties. These consequences are intensified during the school years when children become more involved in social and speaking situations. As a result, children and adolescents who stutter frequently experience peer victimization, social isolation and rejection, and they may also be less popular than their non-stuttering peers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 years to 16 years
* Gender: both sex is included in the study
* Intelligence quotient ≥ 85

Exclusion Criteria:

* Intelligence quotient < 85
* Age below 6 years or above 16 years
* Presence of other speech, language or physical disorders

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Stuttering severity index | 30 minutes
  Score of stuttering severity index a ranging from 1 to 40. It grades was divided into (very mild- mild- moderate- severe- very severe)

SECONDARY OUTCOMES:
Child Behavior Checklist for age 4-18 | 30 minutes
  Questionnaire for detect presence of anxiety in children

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iverach L, Rapee RM. Social anxiety disorder and stuttering: current status and future directions. J Fluency Disord. 2014 Jun;40:69-82. doi: 10.1016/j.jfludis.2013.08.003. Epub 2013 Sep 2. PMID 24929468
- [Background] Smith KA, Iverach L, O'Brian S, Kefalianos E, Reilly S. Anxiety of children and adolescents who stutter: a review. J Fluency Disord. 2014 Jun;40:22-34. doi: 10.1016/j.jfludis.2014.01.003. Epub 2014 Feb 9. PMID 24929464
- [Background] Blood GW, Blood IM, Maloney K, Meyer C, Qualls CD. Anxiety levels in adolescents who stutter. J Commun Disord. 2007 Nov-Dec;40(6):452-69. doi: 10.1016/j.jcomdis.2006.10.005. Epub 2006 Nov 28. PMID 17126361
- [Background] Alm PA. Stuttering in relation to anxiety, temperament, and personality: review and analysis with focus on causality. J Fluency Disord. 2014 Jun;40:5-21. doi: 10.1016/j.jfludis.2014.01.004. Epub 2014 Feb 8. PMID 24929463